CLINICAL TRIAL: NCT01067027
Title: Control of Colic in Infants by Dietary Supplementation With the Probiotic Lactobacillus Reuteri
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Investigational Research Program, LLC (Other)
Responsible Party: Bryan M. Harvey, M.D., Children's Investigational Research Program
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Colic001
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Colic
Keywords: Colic; Colic in Breast-fed Infants
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — 5 drops of study product 30 minutes before feeding.

SUMMARY:
It is believed that probiotic Lactobacillus reuteri will improve the symptoms of breast-fed infants with colic.

ELIGIBILITY:
Inclusion Criteria:

* Ifants aged between 14 and 60 days
* Breast fed, exclusively during length of trial
* Diagnosis of infantile colic according to Wessel's criteria i.e paroxysmal fussing in infancy for more than three hours per day, at least three days per week.
* Debut of colic symptoms 6+/-1 days before randomization
* Gestational age between 37 and 42 weeks
* Apgar score higher than 7 at 5 minutes
* Mothers willing to follow a cows mild-free diet (free from mild, yoghurt, cheese etc) during the study period
* Written informed consent from one or both parents
* Stated availability throughout the study period

Exclusion Criteria:

* Major chronic disease
* Gastrointestinal disease but controlled GERD with or without medication is not an exclusion criteria
* Administration of anitbiotics the week before randomization
* Administration of probiotics the week before randomization
* Participation in other clinical trials

Ages: 14 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
* Reduction of daily average crying time to less than 3 hours from baseline to the end of the study period as measured using a daily reporting of crying time by the parents. | 7, 14 and 21 days

SECONDARY OUTCOMES:
Number of responders versus non-responders with L. reuteri versus placebo at end of the study. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Bryan M Harvey, M.D., Principal Investigator — Children's Investigational Research Program
Locations (1):
- Children's Investigational Research Program, Bentonville, Arkansas, United States